CLINICAL TRIAL: NCT01087190
Title: A Prospective, Randomized, Open Labeled Trial of Isoniazid Treatment Based on ELISPOT Assay to Prevent Tuberculosis in a Kidney Transplant Recipient
Brief Title: Isoniazid (INH) Treatment Based on ELISPOT Assay
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Asan Medical Center (Other)
Responsible Party: Principal Investigator, Sung-Han Kim, Assistant Professor, Asan Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2010-0009
Record Dates: First submitted 2010-03-11; First posted 2010-03-16 (Estimated); Last update posted 2013-12-12 (Estimated); Status verified 2013-12

CONDITIONS: Kidney Transplant Recipient
Keywords: kidney; transplantation; tuberculosis; ELISPOT; isoniazid
MeSH Terms: conditions — Tuberculosis

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- INH treatment group (Experimental): * randomly allocated to INH treatment group in renal transplant recipients with ELISPOT (+)
  * INH 300 mg po qd for 9 months
  Interventions: Drug: Isoniazid treatment
- Control group (No Intervention): * randomly allocated to control group in renal transplant recipients with ELISPOT (+)
  * no treatment
- Observation group (No Intervention): * allocated to observation group in renal transplant recipients with ELISPOT (-)
  * no treatment

INTERVENTIONS:
Drug: Isoniazid treatment — isoniazid 300 mg po qd for 9 months
  Arms: INH treatment group

SUMMARY:
It has been recommended that all transplant recipients undergo a tuberculin skin test (TST) before transplantation. However, the ability of TST to diagnose latent tuberculosis infection (LTBI) in transplant candidates has been reported to be suboptimal because of high rates of false-negative and false-positive results. The enzyme-linked immunospot assay (ELISPOT) detecting interferon-gamma secreting T-cells for diagnosing tuberculosis infection gave promising results in immunocompromised patients as well as in immunocompetent patients. The investigators will perform a randomized, open-label, prospective trial of isoniazid (INH) prophylaxis based on ELISPOT assay for LTBI in renal transplant recipients.

DETAILED DESCRIPTION:
Our previous data have shown that ELISPOT assay was more sensitive to detect LTBI in renal transplant recipients than TST (Kim SH, et al. Transplant Infect Dis 2010 Jan 25 [Epub ahead of print]). However, further studies are eagerly awaited to determine the efficacy of isoniazid (INH) prophylaxis based on ELISPOT assay for LTBI in renal transplant recipients. All adult patients admitted for renal transplantation between May 2010 and April 2013 at the Asan Medical Center, Seoul, South Korea, will be prospectively enrolled. INH (300 mg/day for 9 months) prophylaxis group and no prophylaxis group (control group) will be randomly assigned to all patients with a baseline positive ELISPOT assay regardless of the results of TST. The investigators will compare cumulative probability of developing active TB after transplantation between INH prophylaxis group and control group as primary outcome. Secondary outcomes will be adverse drug reactions, rejection episodes, graft survival, and mortality.

ELIGIBILITY:
Inclusion Criteria:

* 16 years or more
* Kidney transplant recipients

Exclusion Criteria:

* Patients who do not receive isoniazid treatment due to abnormal liver function (i.e. Child-Pugh Score B or C)
* Patients who have clinical risk factors for latent tuberculosis infection

  1. Close contact with a person with pulmonary TB within the past year
  2. Abnormal chest radiography and no prior prophylaxis
  3. A history of untreated or inadequately treated TB
  4. New infection (i.e. a recent conversion of TST to positive status)

     * If kidney transplant donor has these clinical risk factors for latent tuberculosis infection, the transplant recipient from this donor will be excluded from this study.

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 831 (Actual)
Dates: Start 2010-06; Primary Completion 2013-05 (Actual); Study Completion 2013-11 (Actual)

PRIMARY OUTCOMES:
Development of tuberculosis (the rate of tuberculosis after transplantation) | 3 years
  Confirmed tuberculosis Probable tuberculosis Suspected or possible tuberculosis

SECONDARY OUTCOMES:
All cause deaths | 3 years
  * TB-associated deaths
  * non-TB-associated deaths
INH-associated adverse drug reactions | 3 years
  liver function abnormalities
Graft failure | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Sung-Han Kim, MD, Principal Investigator — Asan Medical Center
Locations (1):
- Asan Medical Center, Seoul, South Korea